CLINICAL TRIAL: NCT01275638
Title: The Effect of Moderate-Dose Steroid Therapy in Sepsis: A Placebo-Controlled, Randomized Study
Brief Title: The Effect of Moderate-Dose Steroid Therapy in Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: TC Erciyes University, Erciyes University Medical Faculty
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03/05
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2005-04

CONDITIONS: Sepsis
Keywords: cortisol, prednisolone, adrenal insufficiency, sepsis
MeSH Terms: conditions — Sepsis; Adrenal Insufficiency | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prednisolone (20 mg/day) for 10 days. (Placebo Comparator)
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Prednisolone — Soon after the presumptive diagnosis of severe sepsis, initial laboratory specimens were obtained within 2 hours, and the patients were randomized to treatment with prednisolone or placebo groups. The treatment groups were determined by a computer-generated randomization procedure (in a 1:1 ratio). The steroid group received prednisolone at a moderate-dose (20 mg/day). Prednisolone was given intravenously at 06.00 (10 mg) 14.00 (5 mg) and 22.00 (5 mg) for 10 days. The standard therapy group received a placebo infusion containing physiological saline solution in an identical manner. Patients and their primary physicians were blinded as to which therapy was administered.
  Other Names: prednisolon; prednizolone

SUMMARY:
Despite the new developments in sepsis treatment, mortality rate is still high. Discussions on steroid treatment in sepsis are going on. In this study, we aimed to investigate the effects of moderate dosage steroid treatment and endocrinologic changes occurring in sepsis on prognosis in patients with sepsis.

DETAILED DESCRIPTION:
This prospective, randomized, single-centre, double-blind, placebo-controlled trial was conducted between April 2005 and May 2008 in the department of Medical ICU and the Department of Infectious Diseases of Erciyes University Medical School. The study was approved by our Institutional Review Board and informed consent was obtained from the patients' relatives. The study did not alter therapy, and each patient's clinical care was determined by their own physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 17 years old and diagnosed with sepsis were included in the study consecutively

Exclusion Criteria:

* Already known pre-existing adrenal disease or adrenalectomy, known malignancies, tuberculosis that might have involved the adrenal gland, and administration of steroids within the 3 months before the admission. In addition, patients with burns, hemorrhagic shock or those who had suffered myocardial infarction were not included.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 28-day

SECONDARY OUTCOMES:
Adverse Events | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bilgehan AYGEN, Prof., Study Chair — Erciyes University Medical Faculty Infectious Diseases Departmen